CLINICAL TRIAL: NCT01976624
Title: Safety and Efficacy of Bimatoprost/Timolol (Ganfort®) Ophthalmic Solution in Korea
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 192024-087
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Results first posted 2015-07-21 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-08

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost; Timolol; Ganfort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ganfort®: Patients who received treatment with bimatoprost/timolol (Ganfort®) for open-angle glaucoma or ocular hypertension as per local standard of care in clinical practice.
  Interventions: Drug: bimatoprost/timolol

INTERVENTIONS:
Drug: bimatoprost/timolol — Bimatoprost/timolol (Ganfort®) treatment for open-angle glaucoma or ocular hypertension as per local standard of care in clinical practice.
  Other Names: Ganfort®

SUMMARY:
This study is a Post-Marketing Surveillance study to evaluate the safety and efficacy of bimatoprost/timolol (Ganfort®) Ophthalmic Solution to treat open-angle glaucoma or ocular hypertension in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with Ganfort® for open-angle glaucoma or ocular hypertension in clinical practice.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with Ganfort® for open-angle glaucoma or ocular hypertension in clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 756 (Actual)
Dates: Start 2009-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ganfort®
Started | 756
Completed | 742
Not Completed | 14
Not completed — Participants contraindicated | 2
Not completed — Participants age less than 19 years | 12

BASELINE CHARACTERISTICS:
Population: Safety population included all participants treated for on-label indications.
Arm/Group | Ganfort®
Number analyzed (Participants) | 742
Age, Customized [Number; unit: participants]
  18 to <30 years | 23
  30 to 39 years | 67
  40 to 49 years | 91
  50 to 59 years | 167
  60 to 69 years | 196
  70 to 79 years | 151
  ≥80 years | 46
  Data not Available | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 316
  Male | 426

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events and Adverse Drug Reactions
Description: An Adverse Event was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. An Adverse Drug Reaction was a harmful and unintended reaction that is incurred during routine administration or use of the drug, whose causal relationship with the drug cannot be excluded.
Time Frame: Up to 51 months
Population: Safety population included all participants treated for on-label indications.
Measure: Number; unit: participants
Arm/Group | Ganfort®
Number analyzed (Participants) | 742
participants
  Adverse Events | 146
  Adverse Drug Reactions | 134

2. Secondary Outcome: Change From Baseline in Intraocular Pressure (IOP)
Description: IOP is a measurement of the fluid pressure inside the eye. A negative change from Baseline indicated an improvement. The median total treatment duration for participants was 63.0 days.
Time Frame: Baseline, Week 4
Population: Efficacy population included all participants who were treated for on-label indications with data available for analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ganfort®
Number analyzed (Participants) | 641
mmHg
  Right Eye: Baseline (n=608) | 18.23 (6.69)
  Right Eye: Change from Baseline (n=608) | -3.28 (5.32)
  Left Eye: Baseline (n=616) | 18.23 (6.48)
  Left Eye: Change from Baseline (n=616) | -3.50 (5.24)

ADVERSE EVENTS:
Description: The Safety Population, all participants treated for on-label indications, was used to determine the number of participants at risk for Serious Adverse Events and Adverse Events.
Arm/Group | Ganfort®
Serious Adverse Events (participants affected / at risk) | 1/742
Other Adverse Events (participants affected / at risk) | 86/742
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ganfort® (N=742)
Neoplasm metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Investigator determined not-related to study medication.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ganfort® (N=742)
Conjunctival hyperaemia (Eye disorders) | 86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is at least 30 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.